CLINICAL TRIAL: NCT03487484
Title: Quality of Life in Patients With Rectal Cancer Receiving Neoadjuvant Chemotherapy, Total Mesorectal Excision With or Without Stoma and Adjuvant Chemotherapy: a Prospective, Single-centre Pilot-study
Brief Title: Quality of Life in Patients With Rectal Cancer Receiving Total Mesorectal Excision With or Without Stoma
Status: Terminated | Type: Observational
Why Stopped: insufficient recruitment
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: QoL Rectal Cancer
Record Dates: First submitted 2018-03-26; First posted 2018-04-04 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With protective stoma: Patients in which intraoperatively the decision was made to add a protective stoma (following a risk algorithm) to total mesorectal excision. In patients quality of life, the Gastrointestinal Quality of Life Index (GIQLI) questionnaire, Quality of Life Questionnaire for gastrointestinal tract and Faecal Incontinence Score will be applied.
  Interventions: Behavioral: Quality of Life Questionnaire for gastrointestinal tract; Behavioral: Quality of Life Questionnaire; Behavioral: Faecal Incontinence Score
- No stoma: Patients in which intraoperatively the decision was made to refrain from adding a protective stoma (following a risk algorithm) to total mesorectal excision.
  In patients quality of life, the GIQLI questionnaire (Gastrointestinal Quality of Life Index), Quality of Life Questionnaire for gastrointestinal tract and Faecal Incontinence Score will be applied.
  Interventions: Behavioral: Quality of Life Questionnaire for gastrointestinal tract; Behavioral: Quality of Life Questionnaire; Behavioral: Faecal Incontinence Score

INTERVENTIONS:
Behavioral: Quality of Life Questionnaire for gastrointestinal tract — To assess quality of life, the GIQLI questionnaire (Gastrointestinal Quality of Life Index) will be applied
  Other Names: GIQLI questionnaire
Behavioral: Quality of Life Questionnaire — To assess quality of life, the SF-36 questionnaire will be applied
  Other Names: SF-36 questionnaire
Behavioral: Faecal Incontinence Score — To assess faecal incontinence, the Vaizey Wexner questionnaire will be applied
  Other Names: Vaizey Wexner questionnaire

SUMMARY:
The goal is to evaluate whether the renunciation of a diverting stoma in patients with adjuvant chemotherapy after low anterior resection with total mesorectal excision (TME) and neoadjuvant chemoradiotherapy leads to a better quality of life without increasing morbidity and mortality in patients with rectal cancer.

DETAILED DESCRIPTION:
In most cases it is recommended that patients after low anterior resection with TME and neoadjuvant chemoradiotherapy for rectal cancer need a temporarily diverting stoma. Recent evidence suggests that this is not always necessary. The decision for or against a stoma is made by the surgeon in charge and is based on an algorithm of risk factors for anastomotic leakage. Many patients receive an adjuvant chemotherapy postoperative. This may influence the quality of life e.a. due to mucositis and urge incontinency or the stoma itself.The objective of this pilot study is to establish the basis for a randomized controlled trial. The long-term goal is to evaluate whether the renunciation of a diverting stoma in patients with adjuvant chemotherapy after low anterior resection with TME and neoadjuvant chemoradiotherapy leads to a better quality of life without increasing morbidity and mortality in patients with rectal cancer. All patients scheduled for low anterior resection of the rectum for rectal carcinoma will be invited to participate and prospectively enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

* age older than 18,
* low anterior resection and TME due to rectum carcinoma after standardized neoadjuvant combined chemo- and radiotherapy and receiving adjuvant postoperative chemotherapy,
* German speaking patient who is capable to fill in the questionnaire,
* signed informed consent

Exclusion Criteria:

* age younger than 18,
* preoperative stoma,
* not German speaking
* inability to fill in the questionnaire,
* no standardized chemo- and radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed rectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2020-03-22 (Actual); Study Completion 2020-03-22 (Actual)

PRIMARY OUTCOMES:
Change in quality of life specific for the gastrointestinal tract | at Baseline and up to 12 months after surgery
  GIQLI Score

SECONDARY OUTCOMES:
Change in quality of life | at Baseline and up to 12 months after surgery
  Short Form (SF) 36
Change in faecal Incontinence | at Baseline and up to 12 months after surgery
  Vaizey Wexner Score

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Drews, MD, Principal Investigator — Claraspital Basel
Locations (1):
- St Claraspital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No